CLINICAL TRIAL: NCT05922345
Title: A Multicenter, Randomized, Double-blind, Parallel-controlled Phase III Clinical Trial to Evaluate the Efficacy and Safety of AL2846 Capsules Combined With TQB2450 Injection Compared With Docetaxel Injection in Patients With Advanced Non-small Cell Lung Cancer Who Have Failed With Immunotherapy.
Brief Title: Evaluation of the Efficacy and Safety of AL2846 Capsule Combined With TQB2450 Injection Compared to Docetaxel Injection in Advanced Non-small Cell Lung Cancer Patients Who Have Failed With Immunotherapy.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQB2450-AL2846-III-01
Record Dates: First submitted 2023-06-06; First posted 2023-06-28 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-06

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB2450 injection + docetaxel injection matching placebo + AL2846 capsules (Experimental): TQB2450 injection combined with docetaxel injection matching placebo and AL2846 capsules 21 days as a treatment cycle.
  Interventions: Drug: TQB2450 injection, docetaxel injection matching placebo, AL2846 capsules
- TQB2450 placebo + docetaxel injection + AL2846 placebo (Active Comparator): TQB2450 placebo combined with docetaxel injection and AL2846 placebo 21 days as a treatment cycle.
  Interventions: Drug: TQB2450 placebo, docetaxel injection, AL2846 matching placebo

INTERVENTIONS:
Drug: TQB2450 injection, docetaxel injection matching placebo, AL2846 capsules — AL2846 capsules is a multi-targeted small molecule receptor tyrosine kinase inhibitor.
  TQB2450 Injection is an anti-programmed death-1 (PD-L1).
  Arms: TQB2450 injection + docetaxel injection matching placebo + AL2846 capsules
Drug: TQB2450 placebo, docetaxel injection, AL2846 matching placebo — Docetaxel injection is a type of chemotherapy for treatment of different types of cancer.
  Arms: TQB2450 placebo + docetaxel injection + AL2846 placebo

SUMMARY:
To investigate the efficacy of AL2846 capsules in combination with TQB2450 injection or Docetaxel injection in patients with advanced NSCLC who have previously failed immune checkpoint inhibitors (anti-PD-1 monoclonal antibody, anti-PD-L1 monoclonal antibody), regardless of new anti-tumor treatment and early termination of treatment.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily joined the study, signed an informed consent form, and had good compliance
* Age: 18-75 years; Eastern Eastern Cooperative Oncology Group performance status (ECOG PS) score: 0-1; BMI ≥ 17 at baseline;
* Patients with histologically or cytologically confirmed inoperable and inoperable locally advanced (stage IIIB/IIIC), metastatic or recurrent (stage IV) nonsmall-cell lung cancer (NSCLC) who cannot receive radical concurrent chemoradiotherapy;
* Failure of platinum-based chemotherapy and immune checkpoint inhibitors for incurable locally advanced or metastatic or recurrent NSCLC;
* Number of lines of prior systemic therapy received for locally advanced or metastatic/recurrent disease that is unresectable/not amenable to radical chemoradiation;
* Confirmed to have at least one measurable lesion according to Response Evaluation Criteria In Solid Tumours（ RECIST 1.1） standard;
* Adequate major organ function;

Exclusion Criteria:

* Patients who Have been diagnosed or currently had other malignant tumors;
* Presence of epidermal growth factor receptor (EGFR) mutation, anaplastic lymphoma kinase (ALK) fusion, c-ros oncogene 1 (ROS1) fusion and other significant driver gene mutations;
* Factors affecting oral drugs;
* Major surgical treatment, incisional biopsy or obvious traumatic injury and long-term uncured wound or fracture within 28 days before the start of study treatment;
* Hyperactive/venous thrombotic events within 6 months;
* Subjects with any severe and/or uncontrolled disease;
* Previously received other immunotherapy and Research Advance of Small Molecular Targeted Anti-Tumor Agents Tyrosine kinase inhibitors (TKIs);
* According to the investigator's judgment, there are concomitant diseases that seriously endanger the subject's safety or affect the completion of the study, or there are other reasons that are not suitable for the subject;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From randomization to the time of death from any cause, assessed up to 36 months.
  The time from randomization to the date of death from any cause.

SECONDARY OUTCOMES:
Progression-free survival (PFS) by investigator assessment | From the date of randomization to the date of first recorded progression or death from any cause, whichever comes first, assessed up to 36 months.
  Time from randomization to objective disease progression or death from any cause, whichever occurs first.
Objective response rate (ORR) | Time from the date of randomization to the first recorded complete remission (CR) or partial remission (PR), assessed up to 36 months.
  Refers to the percentage of subjects with complete response (CR) or partial response (PR) as determined by the investigator according to Response Evaluation Criteria in Solid Tumours (RECIST) 1.1.
Disease Control Rate (DCR) | Time from randomization date to CR, PR, or SD or 6 weeks, whichever came first.
  Refers to the percentage of subjects with complete response (CR), partial response (PR) or stable disease (SD) ≥ 6 weeks as determined by the investigator according to RECIST 1.1.
Duration of response (DOR) | From the date of first documentation of tumor response to the date of first documentation of disease progression or death due to any cause, whichever occurs first, assessed up to 36 months.
  For subjects with a best response of complete response (CR) or partial response (PR), it is defined as the time from the date of first documentation of tumor response to the date of first documentation of disease progression or death due to any cause, whichever occurs first.
12-month survival rate (12-month OS rate) | Baseline up to 12-month
  The survival curve corresponds to the cumulative survival rate at 12 months
Health Questionnaire Form | During the screening period, the second cycle and other even numbered cycles, each cycle is 21 days, assessed up to 36 months.
  Questionnaire: pain score：Place a check in the space that best reflects patients' health for the day.
Effects on subjects' health-related quality of life | During the screening period, the second cycle and other even numbered cycles, each cycle is 21 days, assessed up to 36 months.
  Questionnaire: Quality of life related scale (The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire 3rd edition).For questions 1 to 28, choose a number from 1 to 4, 1 means none and 4 means very good. For questions 29 and 30, choose a number from 1 to 7, with 1 being very poor and 7 being very good.
Patients with abnormal laboratory inspection indicators | From signing the informed consent form to the 30 days after the last dose.
  Laboratory inspection indicators exceed the normal range
Adverse event rate | From signing the informed consent form to the 30 days after the last dose.
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs).
Occurrence of anti-drug antibody (ADA) | Pre-dose in cycle 1, cycle 2, cycle 5, cycle 9, 90 days after administration, each cycle is 21 days.
  Occurrence of ADA immunoglobulin
Occurrence of neutralizing antibody (Nab) | Pre-dose in cycle 1, cycle 2, cycle 5, cycle 9, 90 days after administration, each cycle is 21 days.
  Antibody preventing cells from being invaded by an antigen or infectious agent.
Peak Concentration (Cmax) | 60 minutes pre-dose on cycle 1 day 1, cycle 2 day 1, cycle 5 day 1, cycle 9 day 1; 10 minutes post dose on cycle 1 day 1, each cycle is 21 days.
  The highest plasma concentration of a drug reached after administration.
Trough concentration (Cmin) | 60 minutes pre-dose on cycle 1 day 1, cycle 2 day 1, cycle 5 day 1, cycle 9 day 1; 10 minutes post dose on cycle 1 day 1, each cycle is 21 days.
  The lowest concentration of a drug at steady state after multiple doses.
Peak time | 60 minutes pre-dose on cycle 1 day 1, cycle 2 day 1, cycle 5 day 1, cycle 9 day 1; 10 minutes post dose on cycle 1 day 1, each cycle is 21 days.
  The time it takes for a drug to reach Cmax.
Area under the drug time curve (AUC) | 60 minutes pre-dose on cycle 1 day 1, cycle 2 day 1, cycle 5 day 1, cycle 9 day 1; 10 minutes post dose on cycle 1 day 1, each cycle is 21 days.
  The area under the curve of drug concentration in blood over time.
Clearance | 60 minutes pre-dose on cycle 1 day 1, cycle 2 day 1, cycle 5 day 1, cycle 9 day 1; 10 minutes post dose on cycle 1 day 1, each cycle is 21 days.
  It represents the amount of drug cleared per unit of time, reflecting the body's ability to dispose of the drug.
Apparent volume of distribution (Vd) | 60 minutes pre-dose on cycle 1 day 1, cycle 2 day 1, cycle 5 day 1, cycle 9 day 1; 10 minutes post dose on cycle 1 day 1, each cycle is 21 days.
  Describes the extent of drug distribution in the body.
The elimination half-life (t1/2) | 60 minutes pre-dose on cycle 1 day 1, cycle 2 day 1, cycle 5 day 1, cycle 9 day 1; 10 minutes post dose on cycle 1 day 1, each cycle is 21 days.
  The time it takes for the drug concentration to drop to half of its original level.

CONTACTS AND LOCATIONS:
Locations (70):
- China (70):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital Capital Medical University, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Chest Hospital Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Three Gorges Hospital Affiliated to Chongqing University, Chongqing, Chongqing Municipality
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - Meizhou People's Hospital, Meizhou, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - Zhongshan City People's Hospital, Zhongshan, Guangdong
  - Guigang people's hospital, Guigang, Guangxi
  - Liuzhou people's hospital, Liuchow, Guangxi
  - Guangxi Medical University Afiliated Tomor Hospital, Nanning, Guangxi
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - The Second Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - The Second Affiliated Hospital of Hainan Medical College, Haikou, Hainan
  - Hainan Provincial People's Hospital, Haikou, Hainan
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Affiliated Hospital of Chengde Medical College, Chengde, Hebei
  - Tangshan People's Hospital, Tangshan, Hebei
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - Affiliated Cancer Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Jiamusi Tuberculosis Hospital (Jiamusi Cancer Hospital), Jiamusi, Heilongjiang
  - Tong Ji Hospital Affiliated To Tongji Medical College HUST, Wuhan, Hubei
  - Hubei Cancer Hospital (HBCH), Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - XuZhou Central Hospital, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shenyang Tenth People'S Hospital, Shenyang, Liaoning
  - The Second Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shaanxi
  - The First Affiliated Hospital of Air Force Medical University, Xi'an, Shaanxi
  - The Second Affiliated Hospital of the Military Medical University of the PLA Air Force, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Heze Municipal Hospital, Heze, Shandong
  - The Second Hospital of Shandong University, Jinan, Shandong
  - Shandong Cancer Hospital&Institute, Jinan, Shandong
  - Affiliated Hospital of Jining Medical Uniwersity, Jining, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Changzhi People'S Hospital, Changzhi, Shanxi
  - Heping Hospital Affiliated to Changzhi Medical College, Changzhi, Shanxi
  - Linfen Central Hospital, Linfen, Shanxi
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - Affiliated Hospital of North SIchuan Medical College, Nanchong, Sichuan
  - The second people's hospital of neijiang, Neijiang, Sichuan
  - TianJin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - Affiliated Tumor Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The First Affliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Taizhou Enze Medical Center (Group), Taizhou, Zhejiang